CLINICAL TRIAL: NCT02292069
Title: Open Label, Randomized, Two-treatment, Two-period, Two-sequence, Oral Bioequivalence Study of Amlodipine Besylate/Atorvastatin Calcium Tablets 10mg/80mg Under Fed Condition
Brief Title: Bioavailability Study of Amlodipine Besylate/Atorvastatin Calcium Tablets 10/80 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-VIN-107
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine; Atorvastatin; amlodipine, atorvastatin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine besylate/Atorvastatin calcium tablets 10/80 mg (Experimental): Amlodipine besylate/Atorvastatin calcium tablets 10/80 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Amlodipine besylate/Atorvastatin calcium
- Caduet (Active Comparator): Caduet® 10/80 mg tablets of Pfizer, Ireland
  Interventions: Drug: Amlodipine besylate/Atorvastatin calcium

INTERVENTIONS:
Drug: Amlodipine besylate/Atorvastatin calcium — Amlodipine besylate/Atorvastatin calcium 10/80 mg
  Other Names: Caduet

SUMMARY:
This study is to assess the bioequivalence between Amlodipine besylate/Atorvastatin calcium Tablets 10mg/80mg of Dr. Reddy's Laboratories Limited, India and CADUET® (amlodipine besylate and atorvastatin calcium) tablets 10mg/80mg of Pfizer Ireland Pharmaceuticals Dublin, Ireland in healthy, adult,human subjects under Fed conditions.

DETAILED DESCRIPTION:
Open label, randomized, two-treatment, two-period, two-sequence, oral bioequivalence study of Amlodipine besylate/Atorvastatin calcium Tablets 10mg/80mg under Fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 years (both inclusive).
2. Subjects' weight within normal range according to normal values for Body Mass Index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable reference range.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (P/A view) whose X-Ray was taken not more than 6 months prior to the dosing of Period 01.
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breath test.
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

1. Hypersensitivity to Amlodipine and Atorvastatin or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of significant alcoholism or drug abuse.
5. History or presence of significant smoking (more than 10 cigarettes or beedi's/day).
6. History or presence of asthma, urticaria or other significant allergic reactions.
7. History or presence of significant gastric and/or duodenal ulceration.
8. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
9. History or presence of cancer.
10. Difficulty with donating blood.
11. Difficulty in swallowing solids like tablets or capsules.
12. Use of any prescribed or OTC medication during last two weeks prior to dosing in period 01.
13. Major illness during 3 months before screening.
14. Participation in a drug research study within past 3 months.
15. Donation of blood in the past 3 months before screening.
16. Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol for within 48 hours prior to dosing.
17. Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
18. History or presence of significant easy bruising or bleeding.
19. History or presence of significant recent trauma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | The post dose samples of 4.0 mL were drawn at 0.50, 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 11.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours for Amlodipine assay

SECONDARY OUTCOMES:
Area under curve (AUC) | post dose samples of 4.0mL were drawn at 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 2.75, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours for Atorvastatin assay

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Gunjan Shah, MD, Principal Investigator — Veeda Clinical Research Pvt. Ltd
Locations (1):
- Veeda Clinical Research Pvt Ltd, Ahmedabad, Gujarat, India